CLINICAL TRIAL: NCT04673981
Title: Neurosensorial Disorder and Pain in Oral Cavity and Oropharynx Cancer Traited Patients
Brief Title: Neurosensorial Disorder and Pain in Oral Cavity and Oropharynx Cancer Traited Patients (OCAPA)
Acronym: OCAPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2020 PHAM DANG; 2020-A00476-33 (Other: ANSM)
Record Dates: First submitted 2020-09-10; First posted 2020-12-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Head Cancer; Neck Cancer; Chronic Pain
Keywords: Hypoesthesia; Allodynia; Orofacial; Neuropathic pain; cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Chronic Pain; Hypesthesia; Hyperalgesia; Neuralgia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient treated for a oral cavity and oropharynx cancer (Experimental): questionnaire and tests to evaluate neuropathic pain
  Interventions: Diagnostic Test: diagnostic tes for neuropathic pain

INTERVENTIONS:
Diagnostic Test: diagnostic tes for neuropathic pain — Thermotest and hot water, cold water (for the oral cavity), Von frey filament and the brush

SUMMARY:
Following preliminary studies carried out in our department on these subject and subjective findings during clinical examinations, it has been shown that pain is a symptom that is rarely reported following treatment. Instead, neurosensory disorders such as hypoesthesia and paresthesia are found.

The objective of the study is to map and qualitatively evaluate neurosensory disorders in patients treated for cancers of the oral cavity and oropharynx.

DETAILED DESCRIPTION:
The protocol, which is done during the usual follow-up consultation of the patient by the maxillo-facial surgeon, is divided into 3 parts:

PART 1: Collection of Data and Consent

* Patient Data:

  * Date of visit and inclusion in the study
  * Patient initials
  * Age
  * Gender (male or female)
  * The weight
  * The size
* Verification of inclusion and non-inclusion criteria:
* General patient history:

  * Patient history
  * Ongoing Treatments
  * Professional activity
* Tumor:

  * Features
  * Location
  * TNM
  * Histological type
* Search for risk factors for peripheral neuropathy
* Check for symptoms of peripheral neuropathy.

PART 2: Collecting Treatment Data

* Operating data:

  * Operation date
  * Type of surgery
  * Duration of surgery
  * Severed sensory nerves
  * Perioperative complications
* On the way out:

  * Adjuvant treatment including radiotherapy and/or chemotherapy.
  * Exit analgesic treatment
  * EN (Numerical Scale)

PART 3: Collection of data related to neurosensory disorders and pain

* Analgesics consumed
* Questionnaire DN4 for each operated area separated according to the curage, lumpectomy and reconstruction if they take place.
* If DN4 positive, completion of the QCD and QEDN questionnaires.
* Clinical examination for sensory disturbances reported on a chart.
* Generic quality of life questionnaire adapted to cancer pathology EORTC QLQC30 and its specific Head and Neck35 add-on module adapted to head and neck cancers.
* Thermotest and hot water, cold water (for the oral cavity)
* HADS Questionnaire
* Catastrophe Questionnaire
* Quantitative sensory testing (QST) for neuropathic patients :

Mechanical neurosensory disorders will be tested with the Von frey filament and the brush.

* Hypoesthesia or mechanical anaesthesia will be sought with the Von Frey filament and the brush.
* Mechanical hypersensitivity, a painful sensation exacerbated by a sharp, non-traumatic object, will be sought with a large calibre Von Frey filament.
* Static Allodynia, felt painful on contact, will be sought at Von Frey's filament.
* Dynamic Allodynia, felt painful when rubbed, will be sought with a wide brush (8 mm) over a distance of several centimetres.

Thermal neurosensory disorders will be sought for the skin with the Thermotest and at the level of the oral cavity with the application of standardised test tubes containing water at 4°C stored in the fridge or hot water at 63°C (the protocol consists of heating water at 4°C in the microwave for 30 seconds to obtain the temperature of 63°C); these examinations will allow the evaluation of thermal allodynia and hypoesthesia.

The examination will cover the entire face, the oral cavity, the cervical region and the area where the reconstruction flaps are taken. The pathological areas identified will be delimited on diagrams previously made with a coding according to the sensations collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for an oral cavity and oropharynx tumor from at least one year and maximum five years.
* Women or men upper 18 years old)
* Patient with full consent, aware and signed
* Patient cover by the French social security system

Exclusion Criteria:

* Patient with mental disorder, psychologic, with a defect of comprehension to agree fully the protocol
* Pregnant women or nursing
* Patients who can't comply with the protocol
* Participation refusal
* Inable full age patient or under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
hypoesthesia on surgical site using a brush and Von Frey Filament | day 0
  The measure is a binary measure (positive or negative)
anaesthesia on surgical site using a brush and Von Frey Filament | day 0
  The measure is a binary measure (positive or negative)
allodynia on surgical site | day 0
  The measure is a binary measure (positive or negative) by clinical examination
Evaluation of the characteristics of the pain by questionnaire DN4 | Day 0
  One standard DN4 with four questions and ten pain characteristics which gave a score from zero to ten points. If DN4 equal or superior of four out of ten the patient seems possible to develop neuropathic pain.
hyperalgesia on surgical site using a brush and Von Frey Filament | Day 0
  The measure is a binary measure (positive or negative)
Evaluation of the characteristics of the pain by questionnaire Neuropathic Pain Symptom Inventory (NPSI) | Day 0
  Twelve questions with a score from zero to ten, zero stands for no pain and ten maximal pain scale. A score is given for burning pain (score out of ten), constriction pain (score out of ten), paroxystic pain (score out of ten), evoked pain (score out of ten), paresthesia (score out of ten) and a total score (out of one hundred)
Evaluation of the characteristics of the pain by questionnaire Brief Pain Inventory | Day 0
  Fifteen questions compose the questionnaire, the first one is a binary answer yes or no, the second one is a schema to localize the pain, thirteen following questions are scaled with a score from zero to ten, zero stands for no pain and ten maximal pain scale

SECONDARY OUTCOMES:
Questionnaire EORTC QLQC30 to assess Quality of life of cancer patients | day 0
  a score is given for each question, Thirty questions with for each question a score from one (not at all), two (a bit), three (enough) to four (a lot). Two last questions are scale from one (really bad) to seven (excellent)
Questionnaire EORTC QLQ-H&N35 to assess Quality of life of head and neck cancer patient | day 0
  a score is given for 34 questions (with for each question a score from one (not at all), two (a bit), three (enough) to four (a lot)), for the last 5 questions there is a binary scale (1 for no answer and 2 for yes).
Quality of life evaluate by the Questionnaire EORTC QLQ-H&N35 | Day 0
  a score is given for 34 questions (with for each question a score from one (not at all), two (a bit), three (enough) to four (a lot)), for the last 5 questions there is a binary scale (1 for no answer and 2 for yes)
Pain Catastrophizing Scale (PCS-CF) to assess the catastrophizing | Day 0
  thirteen questions with for each question a score from zero (not at all), one (a bit), two (moderatly), three (a lot) to four (constantly).
  A score inferior than thirty mark a moderate risk to develop chronic pain. A score superior than thirty mark a high risk to develop chronic pain.
Anxious and depression disorder screening using questionnaire Hospital Anxiety and Depression scale (HAD) | day 0
  Fourteen items scaled from zero to three, seven questions refer to anxiety seven others to depressive dimension Both of them gathered to make a score of twenty-one for maximum

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie PHAM DANG, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France